CLINICAL TRIAL: NCT04454164
Title: Platelet Rich Plasma In Knee Osteoarthritis: A Prospective, Double-Blind Randomized, Placebo Controlled Clinical Trial
Brief Title: Platelet Rich Plasma Injection for Knee Osteoarthritis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ferhat Say (Other)
Responsible Party: Sponsor-Investigator, Ferhat Say, M.D. Associate Professor, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRP2018
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Knee Osteoarthritis; Cartilage Degeneration
Keywords: platelet-rich plasma; placebo; growth factors; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PRP group (Experimental): Intraarticular 5 ml single PRP injection
  Interventions: Biological: PRP
- Saline group (Placebo Comparator): Intraarticular 5 ml single saline injection
  Interventions: Drug: Saline
- Multiple PRP group (Experimental): Intraarticular 3 dose of 5 ml PRP injection (0, 1, 3 month injection)
  Interventions: Biological: PRP
- Multiple saline group (Placebo Comparator): Intraarticular 3 dose of 5 ml saline injection (0, 1, 3 month injection)
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: PRP — platelet rich plasma
  Other Names: platelet rich plasma
  Arms: Multiple PRP group; PRP group
Drug: Saline — serum physiologic
  Other Names: serum physiologic
  Arms: Multiple saline group; Saline group

SUMMARY:
The research questions of this study are;

1. Is platelet rich plasma (PRP) treatment effective in knee osteoarthritis (OA)?
2. What are the indications for PRP treatment?
3. Which patients are the most suitable for the PRP treatment method?
4. How does age, Body Mass Index (BMI), lower extremity mechanical axis angle and OA stages affect the success of the PRP treatment?
5. Is there any advantage of multiple PRP doses?
6. What is the therapeutic effect of placebo?

This study was designed to find answers of these questions.

The hypotheses of this study are; "PRP treatment is more effective than placebo; PRP treatment effectiveness decreases with age and advanced stages of OA; BMI is a factor that negatively affects the treatment effectiveness of the PRP; as the mechanical axis angle of the lower limb increases, it will adversely affect the effectiveness of PRP therapy; multiple dose of PRP affects the effectiveness and duration of PRP as positively compared to single dose of PRP".

The primary purpose of this study; to prove the effectiveness of PRP treatment on knee pain and functions in patients with knee OA by comparing it with the placebo control group. Secondary purposes of this study; to understand the effect of age, BMI, OA grade and lower limb mechanical axis angle on PRP effectiveness. This study, designed as a randomized, double-blind and placebo control group, with a high level of scientific evidence. Thus, it will be scientifically possible to find answers to the investigators research questions and to prove the investigators hypothesis.

DETAILED DESCRIPTION:
The power analysis of this study was calculated based on the sample size studies of previous studies. The difference of d = 3 units between the two means is to have a standard deviation of 6 units. The sample size 200 required to detect with 95% power in the 95% confidence interval to detect.

This study covers 324 patients. All patients were selected according to predefined and established inclusion and exclusion criteria.

Inclusion criteria were: stage 1-2-3 symptomatic OA patients according to Kellgren / Lawrence staging, age between 18 and 80 years, mean Visual Analogue Score (VAS) of >4 of 10 (worst possible pain) over the course of 7 days during the previous month were included on a voluntary basis. Only one knee injection was made to the patients.

Exclusion criteria were OA secondary to joint inflammatory diseases; patients with generalized OA, metabolic diseases of the bone, coexisting backache, the presence of hematological disease (coagulopathy), bilateral symptomatic lesions and advanced stages (grade 4) of OA; patients who had received intra-articular injections within three months or arthroscopic lavage in the previous one year or who were receiving immunosuppressive; patients with current use of anticoagulant medications or NSAIDs used in the five days before blood donation, major axis deviation (more than 15 degree of varus or more than 5 degree of valgus deviation); and patients with a hemoglobin level less than 11.5 g/dL and platelets level less than 100,000/μL or associated co-morbidities, infection, tumor, crystal arthropathies, anemia, tense joint effusion and pregnancy or possibility of pregnancy.

The voluntary patients included in this study were divided into four different groups with a computer-assisted randomization program. This groups; group A (n:67) were given a single injection of PRP, group B (n:69) were given a single injection of normal saline (physiological control/placebo), group C (n:66) were given three injection (one per month) of PRP, group D (n:65) were given three injection of normal saline (one per month) (physiological control/placebo).

All patients were evaluated by a blinded researcher with VAS, Knee injury and Osteoarthritis Outcome Score (KOOS), Western Ontario and McMaster Universities Arthritis Index (WOMAC), KUJALA, knee range of motion (ROM) and knee circumference measurement at 1st, 3rd, 6th, 12th and 24th months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* stage 1-2-3 symptomatic OA patients according to Kellgren / Lawrence staging
* mean VAS pain score of >4 of 10 (worst possible pain) over the course of 7 days during the previous month

Exclusion Criteria:

* OA secondary to joint inflammatory diseases,
* generalized OA,
* metabolic diseases of the bone,
* coexisting backache,
* the presence of hematological disease (coagulopathy),
* bilateral symptomatic lesions and advanced stages (grade 4) of OA,
* patients who had received intra-articular injections within 3 months or arthroscopic lavage in the previous 1 year,
* patients who were receiving immunosuppressive,
* patients with current use of anticoagulant medications,
* NSAIDs used in the 5 days before blood donation,
* major axis deviation (more than 15 degree of varus or more than 5 degree of valgus deviation),
* patients with a hemoglobin level less than 11.5 g/dL,
* platelets level less than 100,000/μL,
* associated comorbidities, infection, tumor, crystal arthropathies, anemia, tense joint effusion and pregnancy or possibility of pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
VAS | Baseline VAS score
  Visual Analogue scale (0-10 higher scores mean a worse outcome)
VAS | VAS score at 1st months
  Visual Analogue scale (0-10 higher scores mean a worse outcome)
VAS | VAS score at 3th months
  Visual Analogue scale (0-10 higher scores mean a worse outcome)
VAS | VAS score at 6th months
  Visual Analogue scale (0-10 higher scores mean a worse outcome)
VAS | VAS score at 12th months
  Visual Analogue scale (0-10 higher scores mean a worse outcome)
VAS | VAS score at 24th months
  Visual Analogue scale (0-10 higher scores mean a worse outcome)
KOOS | Baseline KOOS score
  Knee injury and Osteoarthritis Outcome Score (0-100 higher scores mean a better outcome)
KOOS | KOOS score at 1st months
  Knee injury and Osteoarthritis Outcome Score (0-100 higher scores mean a better outcome)
KOOS | KOOS score at 3th months
  Knee injury and Osteoarthritis Outcome Score (0-100 higher scores mean a better outcome)
KOOS | KOOS score at 6th months
  Knee injury and Osteoarthritis Outcome Score (0-100 higher scores mean a better outcome)
KOOS | KOOS score at 12th months
  Knee injury and Osteoarthritis Outcome Score (0-100 higher scores mean a better outcome)
KOOS | KOOS score at 24th months
  Knee injury and Osteoarthritis Outcome Score (0-100 higher scores mean a better outcome)
WOMAC | Baseline WOMAC score
  Western Ontario and McMaster Universities Arthritis Index (0-100 higher scores mean a better outcome)
WOMAC | WOMAC score at 1st months
  Western Ontario and McMaster Universities Arthritis Index (0-100 higher scores mean a better outcome)
WOMAC | WOMAC score at 3th months
  Western Ontario and McMaster Universities Arthritis Index (0-100 higher scores mean a better outcome)
WOMAC | WOMAC score at 6th months
  Western Ontario and McMaster Universities Arthritis Index (0-100 higher scores mean a better outcome)
WOMAC | WOMAC score at 12th months
  Western Ontario and McMaster Universities Arthritis Index (0-100 higher scores mean a better outcome)
WOMAC | WOMAC score at 24th months
  Western Ontario and McMaster Universities Arthritis Index (0-100 higher scores mean a better outcome)
Kujala | Baseline Kujala score
  Kujala Patellofemoral Score (0-100 higher scores mean a better outcome)
Kujala | Kujala score at 1st months
  Kujala Patellofemoral Score (0-100 higher scores mean a better outcome)
Kujala | Kujala score at 3th months
  Kujala Patellofemoral Score (0-100 higher scores mean a better outcome)
Kujala | Kujala score at 6th months
  Kujala Patellofemoral Score (0-100 higher scores mean a better outcome)
Kujala | Kujala score at 12th months
  Kujala Patellofemoral Score (0-100 higher scores mean a better outcome)
Kujala | Kujala score at 24th months
  Kujala Patellofemoral Score (0-100 higher scores mean a better outcome)

SECONDARY OUTCOMES:
Knee movement | 1st, 3rd, 6th, 12th and 24th months
  knee joint range of motion (measured by goniometer as degree)
knee circumference | 1st, 3rd, 6th, 12th and 24th months
  Knee Trans patella circumference
mechanical axis angle | baseline
  angle measured from radiological axes graphs
age | baseline
  age of the patient
stage | baseline
  stage of the osteoarthritis
BMI | baseline
  body mass index
patient global satisfaction | 24 months
  subjective satisfaction level of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedic and Trauma, Faculty of Medicine, Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Lin KY, Yang CC, Hsu CJ, Yeh ML, Renn JH. Intra-articular Injection of Platelet-Rich Plasma Is Superior to Hyaluronic Acid or Saline Solution in the Treatment of Mild to Moderate Knee Osteoarthritis: A Randomized, Double-Blind, Triple-Parallel, Placebo-Controlled Clinical Trial. Arthroscopy. 2019 Jan;35(1):106-117. doi: 10.1016/j.arthro.2018.06.035. PMID 30611335
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Background] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Background] Gormeli G, Gormeli CA, Ataoglu B, Colak C, Aslanturk O, Ertem K. Multiple PRP injections are more effective than single injections and hyaluronic acid in knees with early osteoarthritis: a randomized, double-blind, placebo-controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):958-965. doi: 10.1007/s00167-015-3705-6. Epub 2015 Aug 2. PMID 26233594
- [Background] Di Martino A, Di Matteo B, Papio T, Tentoni F, Selleri F, Cenacchi A, Kon E, Filardo G. Platelet-Rich Plasma Versus Hyaluronic Acid Injections for the Treatment of Knee Osteoarthritis: Results at 5 Years of a Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2019 Feb;47(2):347-354. doi: 10.1177/0363546518814532. Epub 2018 Dec 13. PMID 30545242
- [Background] Filardo G, Di Matteo B, Di Martino A, Merli ML, Cenacchi A, Fornasari P, Marcacci M, Kon E. Platelet-Rich Plasma Intra-articular Knee Injections Show No Superiority Versus Viscosupplementation: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1575-82. doi: 10.1177/0363546515582027. Epub 2015 May 7. PMID 25952818
- [Derived] Yurtbay A, Say F, Cinka H, Ersoy A. Multiple platelet-rich plasma injections are superior to single PRP injections or saline in osteoarthritis of the knee: the 2-year results of a randomized, double-blind, placebo-controlled clinical trial. Arch Orthop Trauma Surg. 2022 Oct;142(10):2755-2768. doi: 10.1007/s00402-021-04230-2. Epub 2021 Oct 27. PMID 34705072